CLINICAL TRIAL: NCT03838484
Title: Effects of Transdermal Nicotine on Response Inhibition to Emotional Cues in Schizophrenia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment challenges due to Covid19.
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Florida (Other)
Responsible Party: Principal Investigator, Alan Lewis, Assistant Professor of Psychiatry and Behavioral Sciences, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 190021; 7K23MH116339 (NIH)
Record Dates: First submitted 2019-02-07; First posted 2019-02-12 (Actual); Results first posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Schizophrenia; Impulsive Behavior
Keywords: Nicotine; Nicotinic acetylcholine receptors; Schizophrenia; Schizoaffective disorder; Healthy control; Impulsive behavior; Aggression; Urgency
MeSH Terms: conditions — Schizophrenia; Impulsive Behavior; Psychotic Disorders; Aggression | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Healthy: placebo first, nicotine last (Experimental): Healthy controls will apply placebo skin patch for up to two hours prior to behavioral and EEG task during the first visit in week 1. After a washout period, they will return and apply a nicotine patch (7 mg/24 hour dose) for up to two hours prior to behavioral and EEG task during the second visit in week 2.
  Interventions: Drug: Nicotine Patch, 7 Mg/24 Hr; Drug: Placebo patch
- Healthy: nicotine first, placebo last (Experimental): Healthy controls will apply nicotine skin patch (7 mg/24 hour dose) for up to two hours prior to behavioral and EEG task during the first visit in week 1. After a washout period, they will return and apply a placebo patch for up to two hours prior to behavioral and EEG task during the second visit in week 2.
  Interventions: Drug: Nicotine Patch, 7 Mg/24 Hr; Drug: Placebo patch
- SCZ: placebo first, nicotine last (Experimental): Subjects with schizophrenia (SCZ) will apply placebo skin patch for up to two hours prior to behavioral and EEG task during the first visit in week 1. After a washout period, they will return and apply a nicotine patch (7 mg/24 hour dose) for up to two hours prior to behavioral and EEG task during the second visit in week 2.
  Interventions: Drug: Nicotine Patch, 7 Mg/24 Hr; Drug: Placebo patch
- SCZ: nicotine first, placebo last (Experimental): Subjects with schizophrenia (SCZ) will apply nicotine skin patch (7 mg/24 hour dose) for up to two hours prior to behavioral and EEG task during the first visit in week 1. After a washout period, they will return and apply a placebo patch for up to two hours prior to behavioral and EEG task during the second visit in week 2.
  Interventions: Drug: Nicotine Patch, 7 Mg/24 Hr; Drug: Placebo patch

INTERVENTIONS:
Drug: Nicotine Patch, 7 Mg/24 Hr — Nicotine patch, 7 mg/24 hour will be applied to the skin.
Drug: Placebo patch — Placebo skin patch will be applied to the skin.

SUMMARY:
The purpose of this study is to test whether nicotine, a drug that activates receptors called nicotinic acetylcholine receptors in the brain, improves the ability to make or withhold responses to faces that are either emotionally neutral or emotionally negative. This study will also test whether the drug affects brain activity while making or withholding responses using electroencephalography. Previous studies in people with schizophrenia have shown that more errors in response to negative emotional cues are related to greater likelihood of impulsive aggressive behavior. Therefore, the aim of this study is to determine whether nicotine might be a new strategy to reduce aggressive behavior. The investigators' goal is 25 individuals with schizophrenia and 25 healthy controls to complete the study at Vanderbilt.

DETAILED DESCRIPTION:
This human laboratory study seeks to test the hypothesis that activation of nicotinic acetylcholine receptors (nAChRs) in the brain will reduce impulsive behavior in response to negative emotional cues as compared to neutral emotional cues. Because impulsive action during negative mood states is strongly correlated with impulsive aggression in both healthy individuals and individuals with schizophrenia (discussed below), the investigators' overarching, long-term goal is to determine whether nAChRs in general as well as specific nAChR subclasses might represent novel treatment targets to reduce impulsive aggressive behavior, a significant public health problem.

Nicotinic acetylcholine receptors are a large family of excitatory, pentameric, ionotropic, ligand-gated ion channels located throughout the brain and the remainder of the body. Their endogenous ligand is acetylcholine, yet this family is defined by their common activation by nicotine. Interestingly, anti-aggressive, or "serenic" effects of nicotine have been demonstrated across a number of animal models, including mice, rats, and non-human primates, and multiple human laboratory studies demonstrate an anti-aggressive effect of nicotine in humans. The investigators' laboratory has also demonstrated that acute administration of nicotine at relatively low doses results in reduction of aggressive behaviors in mouse models. Because nicotine is active at all nAChRs, the investigators explored this mechanism further and found that hippocampal alpha-7 nAChRs were both necessary and sufficient for nicotine's serenic effect. Consistent with these findings, there is substantial evidence in humans that reduction of alpha-7 nAChR signaling enhances aggressive behavior, including in individuals with 15q13.3 microdeletion syndrome, a genetic disorder resulting from the deletion of the region of chromosome 15 containing the gene coding for alpha-7 nAChRs. The investigators have also translated these findings into human clinical populations, finding recently the safety and efficacy of transdermal nicotine to reduce aggression and irritability in young adults with autism spectrum disorder. This work, along with other previous case studies in humans, supports targeting nAChRs using transdermal nicotine to reduce aggressive behaviors.

Urgency is a behavioral construct defined as the tendency to act rashly in the context of strong positive or negative emotion, and explains a large degree of variance in the development of impulsive aggression in subjects with schizophrenia and other populations without psychiatric disorders. In patients with schizophrenia, degree of urgency correlates with structural and functional changes in a neuronal network involving prefrontal cortical and limbic/cognitive control brain regions. A number of previous studies have similarly demonstrated impulsivity in the context of negative emotion, called "negative urgency", correlates with history of aggression, as well as substance use and other risky behaviors. Urgency is a hereditable trait that may be considered an endophenotype of impulsive aggression.

Recent studies in humans have explored the relationship between mood-related impulsivity (i.e. urgency) and aggressive behavior using an Emotional Go/NoGo task. This task measures responding or response withholding to visual stimuli of neutral or emotional (typically negative) valence, and quantifies reaction time and commission/omission errors as a function of stimulus valence. Using an Emotional Go/NoGo task, Krakowski et al. studied healthy controls, patients with schizophrenia with or without a history of violence, and non-psychotic individuals with history of violence. In all groups, emotional valence had a significant effect on error commission. In schizophrenia patients, individuals with history of violence were significantly faster to make an incorrect response to negative stimuli (i.e. not withhold a response) than patients without history of violence, whereas the two groups did not differ in response times to neutral valence stimuli. Other studies have also demonstrated an interaction between emotional valence and impulsive errors in schizophrenia, as well as a relationship between emotional valence, impulsive errors, history of violence, and frontal cortex 5-HT1B receptor binding.

While the investigators' studies in mice suggest a direct effect of nAChR stimulation on aggression through activation of the alpha-7 nAChR and are supported by the results using transdermal nicotine in humans, to the investigators' knowledge no previous studies have directly examined the relationship between pharmacological targeting of nAChRs using transdermal nicotine and effects on impulsivity in the context of emotional cues in humans. The investigators now aim to directly test this hypothesis using an Emotional Go/NoGo task in subjects with schizophrenia and healthy controls to determine whether transdermal nicotine improves impulsive behavior and neural correlates in the context of negative and neutral valence cues. Given the relationship between impulsivity and aggressive behavior, the findings of this proposed study will strongly inform future studies of targeting nAChRs broadly and alpha-7 nAChRs more specifically to identify novel treatments for individuals with severe neuropsychiatric disorders struggling with persistent pathological impulsive aggression.

ELIGIBILITY:
Inclusion Criteria for schizophrenia subjects:

1. Men and women age 18 - 65.
2. Communicative in English.
3. Provide voluntary, written informed consent.
4. Physically healthy by medical history,and ECG examination.
5. BMI > 17.5 and < 45.
6. Diagnosis of schizophrenia (ICD-10 F20) or schizoaffective disorder (ICD-10 F25) confirmed by Structured Clinical Interview for Diagnostic and Statistical Manual (DSM)-V (SCID) or diagnostic interview with a trained clinician.
7. Stable medication regimen over at least the past two weeks, including the use of either an oral or intramuscular administration of an antipsychotic medication. Additionally, subjects may take any prescribed medication aside from a nicotine-containing product as long as it has been regularly taken over the past two weeks, including as-needed ("PRN") medication.
8. Negative urine toxicology and negative urine cotinine (to confirm no recent nicotine use) at screening.
9. Does not meet criteria for substance or alcohol use disorder per the SCID over the past 6 months
10. For females, no longer of child-bearing potential, or agreeing to practice effective contraception during the study (e.g., established use of oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device [IUD] or intrauterine system [IUS]; barrier methods: condom with spermicidal foam/gel/film/cream/suppository or occlusive cap [diaphragm or cervical/vault caps] with spermicidal foam/gel/film/cream/suppository; male partner sterilization; or true abstinence when this is in line with the preferred and usual lifestyle of the subject); and,
11. For females of child-bearing potential, must have negative urine pregnancy test at time of screening visit and before each testing day.
12. Not breastfeeding/nursing at time of screening or at any time during the study.

Exclusion Criteria for schizophrenia subjects:

1. Age less than 18 or greater than 65.
2. Not communicative in English.
3. Unable to provide written informed consent.
4. Active suicidal ideation or suicidal behavior.
5. Current, unstable medical or neurological illness or significant abnormality on ECG.
6. History of severe head trauma.
7. BMI < 17.5 or > 45.
8. History of allergy to transdermal patches.
9. Screening visit resting heart rate > 110 or < 50 beats per minute, or known history of clinically significant cardiac rhythm abnormalities.
10. Screening visit systolic blood pressure > 160 or < 90, or diastolic blood pressure > 95 or < 50.
11. Positive urine toxicology or positive urine cotinine during screening.
12. Meets criteria for diagnosis of substance or alcohol use disorder by SCID within the past 6 months.
13. Reports any tobacco smoking or nicotine use over the past month.
14. Not taking an antipsychotic medication.
15. Positive urine pregnancy test at time of screening, before each testing day, or any potential concern for pregnancy at any time during the study
16. Breastfeeding/nursing at time of screening or at any time during the study.

Inclusion Criteria for healthy volunteer subjects:

All of the above except for subjects will be psychiatrically healthy and not taking psychotropic or potentially psychoactive prescription medication.

Exclusion Criteria for healthy volunteer subjects:

All of the above and in addition:

1. Current use of psychotropic or potentially psychoactive prescription medication.
2. Major psychiatric disorder as determined by DSM-5 (schizophrenia, major depression, bipolar disorder, obsessive-compulsive disorder, post-traumatic stress disorder, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan S Lewis, MD, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Psychiatric Hospital, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krakowski MI, De Sanctis P, Foxe JJ, Hoptman MJ, Nolan K, Kamiel S, Czobor P. Disturbances in Response Inhibition and Emotional Processing as Potential Pathways to Violence in Schizophrenia: A High-Density Event-Related Potential Study. Schizophr Bull. 2016 Jul;42(4):963-74. doi: 10.1093/schbul/sbw005. Epub 2016 Feb 19. PMID 26895845
- [Background] Egashira K, Matsuo K, Nakashima M, Watanuki T, Harada K, Nakano M, Matsubara T, Takahashi K, Watanabe Y. Blunted brain activation in patients with schizophrenia in response to emotional cognitive inhibition: a functional near-infrared spectroscopy study. Schizophr Res. 2015 Mar;162(1-3):196-204. doi: 10.1016/j.schres.2014.12.038. Epub 2015 Jan 13. PMID 25595654
- [Background] Lewis AS, van Schalkwyk GI, Lopez MO, Volkmar FR, Picciotto MR, Sukhodolsky DG. An Exploratory Trial of Transdermal Nicotine for Aggression and Irritability in Adults with Autism Spectrum Disorder. J Autism Dev Disord. 2018 Aug;48(8):2748-2757. doi: 10.1007/s10803-018-3536-7. PMID 29536216

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant lost to follow-up
Period: Overall Study
Arm/Group | Healthy: Placebo First, Nicotine Last | Healthy: Nicotine First, Placebo Last | SCZ: Placebo First, Nicotine Last | SCZ: Nicotine First, Placebo Last
Started | 5 | 5 | 4 | 4
Completed | 5 | 4 | 4 | 4
Not Completed | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy: Placebo First, Nicotine Last | Healthy: Nicotine First, Placebo Last | SCZ: Placebo First, Nicotine Last | SCZ: Nicotine First, Placebo Last | Total
Number analyzed (Participants) | 5 | 4 | 4 | 4 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (4) | 38 (11) | 33 (15) | 26 (5) | 33 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 1 | 5
  Male | 4 | 2 | 3 | 3 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 3 | 4 | 4 | 4 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 0 | 0 | 3
  White | 2 | 3 | 4 | 4 | 13
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 4 | 4 | 17

OUTCOME MEASURES:

1. Primary Outcome: False Alarm Error Rate
Description: Participants will be shown fearful, sad, angry, and disgust faces (negative valence) and neutral faces performed in 5 blocks (3 emotional blocks with angry/fearful/sad/disgust faces and 2 non-emotional blocks). In each block the subject is instructed on the go/no-go targets and will press a key ("Go") or withhold pressing a key ("NoGo"). The False Alarm Error Rate will be measured by the proportion of incorrect responses.
Time Frame: Week 1
Population: Please note that this outcome measure specifically refers to the specified outcome measure time frame: week 1. Because this is a crossover trial, only a subset of the subjects completed each treatment (placebo or nicotine) during week 1.
Measure: Mean (Standard Error); unit: Proportion of incorrect responses
Groups:
- Healthy: Placebo: Healthy controls will apply placebo skin patch for up to two hours prior to behavioral and EEG task during the first visit in week 1.
- Healthy: Nicotine: Healthy controls will apply nicotine skin patch (7 mg/24 hour dose) for up to two hours prior to behavioral and EEG task during the first visit in week 1.
- SCZ: Placebo: Subjects with schizophrenia (SCZ) will apply placebo skin patch for up to two hours prior to behavioral and EEG task during the first visit in week 1.
- SCZ: Nicotine: Subjects with schizophrenia (SCZ) will apply nicotine skin patch (7 mg/24 hour dose) for up to two hours prior to behavioral and EEG task during the first visit in week 1.
Arm/Group | Healthy: Placebo | Healthy: Nicotine | SCZ: Placebo | SCZ: Nicotine
Number analyzed (Participants) | 5 | 4 | 4 | 4
Proportion of incorrect responses | 0.20 (0.05) | 0.15 (0.07) | 0.11 (0.04) | 0.19 (0.05)

2. Primary Outcome: False Alarm Error Rate
Description: as for outcome 1
Time Frame: Week 2
Population: Please note that this outcome measure specifically refers to the specified outcome measure time frame: week 2. Because this is a crossover trial, only a subset of the subjects completed each treatment (placebo or nicotine) during week 2.
Measure: Mean (Standard Error); unit: Proportion of incorrect responses
Groups:
- Healthy: Nicotine: Healthy controls will apply nicotine patch (7 mg/24 hour dose) for up to two hours prior to behavioral and EEG task during the second visit in week 2.
- Healthy: Placebo: Healthy controls will apply a placebo patch for up to two hours prior to behavioral and EEG task during the second visit in week 2.
- SCZ: Nicotine: Subjects with schizophrenia (SCZ) will apply a nicotine patch (7 mg/24 hour dose) for up to two hours prior to behavioral and EEG task during the second visit in week 2.
- SCZ: Placebo: Subjects with schizophrenia (SCZ) will apply a placebo patch for up to two hours prior to behavioral and EEG task during the second visit in week 2.
Arm/Group | Healthy: Nicotine | Healthy: Placebo | SCZ: Nicotine | SCZ: Placebo
Number analyzed (Participants) | 5 | 4 | 4 | 4
Proportion of incorrect responses | 0.18 (0.03) | 0.13 (0.06) | 0.15 (0.02) | 0.23 (0.04)

3. Primary Outcome: Omission Error Rate
Description: Participants will be shown fearful, sad, angry, and disgust faces (negative valence) and neutral faces performed in 5 blocks (3 emotional blocks with angry/fearful/sad/disgust faces and 2 non-emotional blocks). In each block the subject is instructed on the go/no-go targets and will press a key ("Go") or withhold pressing a key ("NoGo"). The Omission Error Rate will be measured by the proportion of questions asked with a failure to respond.
Time Frame: Week 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Proportion of omitted responses
Arm/Group | Healthy: Placebo | Healthy: Nicotine | SCZ: Placebo | SCZ: Nicotine
Number analyzed (Participants) | 5 | 4 | 4 | 4
Proportion of omitted responses | 0.24 (0.04) | 0.29 (0.06) | 0.44 (0.06) | 0.27 (0.03)

4. Primary Outcome: Omission Error Rate
Description: as for outcome 3
Time Frame: Week 2
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Proportion of omitted responses
Groups:
- Healthy: Nicotine: Healthy controls will apply a nicotine patch (7 mg/24 hour dose) for up to two hours prior to behavioral and EEG task during the second visit in week 2.
Arm/Group | Healthy: Nicotine | Healthy: Placebo | SCZ: Nicotine | SCZ: Placebo
Number analyzed (Participants) | 5 | 4 | 4 | 4
Proportion of omitted responses | 0.29 (0.07) | 0.23 (0.06) | 0.38 (0.10) | 0.30 (0.03)

5. Primary Outcome: Reaction Time for Correct Hits
Description: Time taken from stimulus presentation to button push during Go trials
Time Frame: Week 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Milliseconds
Arm/Group | Healthy: Placebo | Healthy: Nicotine | SCZ: Placebo | SCZ: Nicotine
Number analyzed (Participants) | 5 | 4 | 4 | 4
Milliseconds | 485.09 (16.56) | 491.05 (16.50) | 468.96 (13.49) | 517.05 (4.66)

6. Primary Outcome: Reaction Time for Correct Hits
Description: Time taken from stimulus presentation to button push during Go trials
Time Frame: Week 2
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Milliseconds
Groups:
- SCZ: Placebo: Subjects with schizophrenia (SCZ) will apply placebo patch for up to two hours prior to behavioral and EEG task during the second visit in week 2.
Arm/Group | Healthy: Nicotine | Healthy: Placebo | SCZ: Nicotine | SCZ: Placebo
Number analyzed (Participants) | 5 | 4 | 4 | 4
Milliseconds | 477.54 (15.06) | 511.10 (10.88) | 478.99 (18.36) | 490.67 (24.40)

7. Primary Outcome: Reaction Time for False Alarms
Description: Time taken from stimulus presentation to button push during NoGo trials
Time Frame: Week 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Milliseconds
Arm/Group | Healthy: Placebo | Healthy: Nicotine | SCZ: Placebo | SCZ: Nicotine
Number analyzed (Participants) | 5 | 4 | 4 | 4
Milliseconds | 718.89 (36.52) | 658.20 (40.50) | 813.00 (48.83) | 692.95 (31.27)

8. Primary Outcome: Reaction Time for False Alarms
Description: Time taken from stimulus presentation to button push during NoGo trials
Time Frame: Week 2
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Milliseconds
Arm/Group | Healthy: Nicotine | Healthy: Placebo | SCZ: Nicotine | SCZ: Placebo
Number analyzed (Participants) | 5 | 4 | 4 | 4
Milliseconds | 727.30 (60.81) | 758.12 (69.68) | 769.95 (42.67) | 703.99 (23.82)

ADVERSE EVENTS:
Time Frame: 30 minutes following removal of patch on each session day.
Description: Adverse event information was collected for any untoward or unfavorable medical occurrence in a participant using the Udvalg for Kliniske Undersøgelser (UKU) side effect rating scale autonomic subscale score. Adverse events were collected from the time the consent was signed through participant completion.
Groups:
- Healthy: Placebo: Healthy controls will apply placebo skin patch for up to two hours prior to behavioral and EEG task.
- Healthy: Nicotine: Healthy controls will apply nicotine skin patch (7 mg/24 hour dose) for up to two hours prior to behavioral and EEG task.
- SCZ: Placebo: Subjects with schizophrenia (SCZ) will apply placebo skin patch for up to two hours prior to behavioral and EEG task.
- SCZ: Nicotine: Subjects with schizophrenia (SCZ) will apply nicotine skin patch (7 mg/24 hour dose) for up to two hours prior to behavioral and EEG task.
Arm/Group | Healthy: Placebo | Healthy: Nicotine | SCZ: Placebo | SCZ: Nicotine
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 2/10 | 4/10 | 2/8 | 3/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy: Placebo (N=10) | Healthy: Nicotine (N=10) | SCZ: Placebo (N=8) | SCZ: Nicotine (N=8)
Blurry vision (Eye disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Increased salivation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Increased urination (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Recruitment for this study did not reach its original intended size due to difficulties from the Covid19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-23): https://cdn.clinicaltrials.gov/large-docs/84/NCT03838484/Prot_SAP_004.pdf
  • Informed Consent Form (2019-10-23): https://cdn.clinicaltrials.gov/large-docs/84/NCT03838484/ICF_005.pdf